

Clinical Study to Evaluate the Safety and Efficacy of the SlimShape Device for Abdominal Fat and Circumference Reduction

 Protocol #
 DHF22621
 Rev. Date
 October 8, 2017
 

This document is the property of **Syneron Medical Ltd**. No part of this document may be reproduced, stored in retrieval system, or transmitted in any form or any means, electronic, mechanical, photocopying, recording or otherwise without prior written permission from **Syneron Medical Ltd**.

Title: Clinical Study to Evaluate the Safety and Efficacy of the SlimShape Device for

Abdominal Fat and Circumference Reduction

**Protocol Number:** DHF22621

**Study Type:** Prospective Clinical Study

Date: September 29, 2016

Study Devices: SlimShape

**Sponsor:** Syneron Medical Ltd.

Industrial Zone, Tavor Building

P.O.B. 160 Yokneam Illit,

20692 Israel

**Project Lead:** Ruthie Amir MD

Global Vice President of Clinical & Regulatory Affairs

ruthiea@syneron.com + 972-73-244-2349

### This document contains confidential information.

This study will be performed in accordance with applicable regulatory requirements and Good Clinical Practice (GCP). This clinical investigation will follow the principles outlined by the International Conference on Harmonization (ICH).



Ruthie Amir, M.D.

# Clinical Study to Evaluate the Safety and Efficacy of the SlimShape Device for Abdominal Fat and Circumference Reduction

 Protocol #
 DHF22621
 Rev. Date
 October 8, 2017
 

Date

| Principal Investigator and study site: | |
|---|---|
| Site: | - |
| Principal Investigator's Signature | |
| I, have carefully "Clinical Study to Evaluate the Safety and Efficacy of the Circumference Reduction" and agree that it contaconducting this study safely. I will conduct this study Good Clinical Practices, and local regulatory guidelines within the time designated. I will provide copies of relating to pre-clinical and prior clinical experience suresponsible to me who participate in the study. I wassure that they are adequately informed regarding the lagree to keep records on all subject information (coreturn forms and all other information collected during Health Canada regulations. | e SlimShape Device for Abdominal Fat and ains all the necessary information for y in strict accordance with this protocol, s, and will attempt to complete the study of the protocol and all other information abmitted by the Sponsor to all personne ill discuss this information with them to e study product and conduct of the study ase report forms, shipment and product |
| ACCEPTED AND AGREED: | |
| Investigator's Signature | Date |



# Clinical Study to Evaluate the Safety and Efficacy of the SlimShape Device for Abdominal Fat and Circumference Reduction

Protocol # DHF22621 Rev. Date October 8, 2017 

# **Table of Contents**

| Glossary | _ |
|----------------------------------------------------------------|----|
| Table 1- Study Synopsis | 6 |
| Introduction and rationale | 8 |
| Background | 8 |
| Device Descriptions | 9 |
| Syneron SlimShape Device | 9 |
| Study design overview | 11 |
| Sutdy Objective | 12 |
| Primary Objective | |
| Primary Safety Objective | |
| Secondary Objectives | 12 |
| Primary and Secondary Efficacy Endpoint | 12 |
| Primary Safety Endpoint | 13 |
| Study population | 13 |
| Number of Subjects | |
| Subject Withdrawal and Replacement | 13 |
| Inclusion Criteria | 13 |
| Exclusion Criteria | 14 |
| STUDY PROCEDURES | 15 |
| Enrollment and Screening | 15 |
| Table 2 – Clinical Evaluation Measurements and Tools | 16 |
| Pre-Treatment Procedures | 17 |
| Screening | 17 |
| Baseline | 17 |
| Measurements | 18 |
| Treatment Procedure | 21 |
| SlimShape Treatment Procedure | 22 |
| Post Treatment Procedures | 24 |
| Return Visits | 24 |
| DATA ANALYSIS | 25 |
| Recording | 25 |
| Demography and Baseline Measurements | 25 |
| Treatment Visit | 25 |
| Follow-up Visit Measurements | 25 |
| Safety | 25 |
| Protocol Revisions and/or Deviations | 25 |
| ADVERSE EVENTS (AE) | |
| Anticipated Adverse Effects | 26 |
| Unanticipated Adverse Device Effects | |
| Reporting Adverse Events (AE) and Serious Adverse Events (SAE) | 27 |



# Clinical Study to Evaluate the Safety and Efficacy of the SlimShape Device for Abdominal Fat and Circumference Reduction

| Measures taken to protect the rights and welfare of subject | 28 |
|----------------------------------------------------------------|----|
| RISK/BENEFIT ANALYSIS | 28 |
| Risks | 28 |
| Potential benefits to participating individuals and to society | 28 |
| Conclusion: | 29 |
| ETHICS AND GOOD CLINICAL PRACTICE | 29 |
| QUALITY ASSURANCE AND STUDY MONITORING | 29 |
| Study Monitoring/Auditing/Inspection | 29 |
| ADMINISTRATIVE PROCEDURES | 30 |
| Supply and Disposition of Study Device | 30 |
| Control & Disposition of the Investigational Device | 30 |
| Informed Consent | 30 |
| Monitoring Plan | 31 |
| Case Report Forms | 31 |
| Record Maintenance | 31 |
| PUBLICATION POLICY | 32 |
| BIBLIOGRAPHY | 33 |
| Appendix I – Study Summery | 34 |
| Appendix II - Scales | 36 |
| Appendix III - Photography | 37 |
| Specific photography details: | 37 |
| Abdomen: | 37 |
| Appendix IV - Clinical Trial Acknowledgement | 38 |



Clinical Study to Evaluate the Safety and Efficacy of the SlimShape Device for Abdominal Fat and Circumference Reduction

Syneron Medical Ltd. Confidential

Protocol # DHF22621 Rev. Date October 8, 2017 

#### **GLOSSARY**

ADE Adverse Device Effect

AE Adverse Event
BMI Body Mass Index

CFR Code of Federal Regulations

Cm Centimeter

CRF Case Report Form

FDA Food & Drug Administration

FU Follow-up

GCP Good Clinical Practice
ICF Informed Consent Form

IEC Institutional Ethics Committee IRB Institutional Review Board

Kg Kilogram Min Minute wk Weeks

PI Principal Investigator

USAE Unanticipated, serious adverse event

USADE Unanticipated, serious adverse device effect

SAE Serious Adverse Event

Tx Treatment US Ultrasound

USI Ultrasound Imaging

W Watt (Output Electric Power)

| Clinical Study to Evaluate the Safety and Efficacy of the SlimShape Device for Abdominal Fat |
|---|
| and Circumference Reduction |

# **TABLE 1- STUDY SYNOPSIS**

| Proprietary Name | SlimShape device |
|---|---|
| Design | Prospective, one arm, baseline-controlled, clinical study for the evaluation of the SlimShape |
| | device for non-invasive abdominal fat and circumference reduction. |
| | Study subjects will undergo SlimShape treatments on the abdominal area |
| Study Population | Up to 120 healthy adult volunteers, seeking for noninvasive abdominal fat and circumference |
| | reduction, male and females, 18 to 60 years of age from up to 10 investigational sites. |
| Treatment and | Eligible subjects will receive up to 3 bi-weekly treatments (2 weeks interval) with the |
| Duration | SlimShape device utilizing the SlimShape Applicator Belt according to the study protocol. |
| | The subject will return for 3 follow up visits: four weeks (4wk FU), eight weeks (8wk FU) and |
| | 12 weeks (12wk FU) after the last treatment. |
| | Each subject will be enrolled for total expected study duration of up to 16 weeks. |
| Objective | The objective of this trial is to evaluate the safety and efficacy of the SlimShape device |
| | utilizing the SlimShape Applicator Belt for abdominal non-invasive fat and circumference |
| | reduction |
| Primary Objective | Statistically significant abdominal fat reduction post SlimShape treatments at 12 weeks |
| | follow-up (12wk FU) versus baseline |
| Primary Safety | Evaluate the safety of the treatment with the SlimShape device utilizing the SlimShape |
| Objective | Applicator Belt during all study |
| Secondary | 1. Statistically significant abdominal fat reduction post SlimShape treatments as |
| Objectives | measured by Ultrasound device at Pre Tx.3, 4 weeks, and 8 weeks follow-up (4wk FU and 8wk FU) versus baseline |
| | Statistically significant abdominal fat reduction post SlimShape treatments as |
| | measured by calibrated Caliper device at Pre Tx.3, 4 weeks, 8 weeks and 12 weeks |
| | follow-up (4wk FU, 8wk FU and 12wk FU) versus baseline |
| | 3. Statistically significant abdominal circumference reduction post SlimShape |
| | treatment/s at Pre Tx.2, Pre Tx.3, 4 weeks, 8 weeks and 12 weeks follow-up (4wk FU, |
| | 8wk FU and 12wk FU) versus baseline |
| | · |
| | 4. Investigator satisfaction: |
| | Satisfaction assessment will be performed by the study investigator using a pre- |
| | defined scale questionnaire. The investigator will answer this questionnaire at each |
| | follow-up visit (4wk FU, 8wk FU and 12wk FU) |

| SYNERON © CANDELA | Clinical Study to Evaluate the Safety and Efficacy of the SlimShape Device for Abdominal Fat and Circumference Reduction | | | | |
|---|---|---|---|---|---|
| Syneron Medical Ltd.<br>Confidential | Protocol # | DHF22621 | Rev. Date | October 8, 2017 | Page <b>7</b> of <b>39</b> |
| | Improveme | provement and satisfacted and satisfaction assing a pre-defined sca | sessment will | • | |

questionnaire at each follow-up visit (4wk FU, 8wk FU and 12wk FU)

| SYNERON O CANDELA' | Clinical Study to Evaluate the Safety and Efficacy of the SlimShape Device for Abdominal Fat and Circumference Reduction | | | | |
|---|---|---|---|---|---|
| Syneron Medical Ltd.<br>Confidential | Protocol # | DHF22621 | Rev. Date | October 8, 2017 | Page <b>8</b> of <b>39</b> |

| Efficacy Endpoints | Primary and secondary objectives will be measured using the next efficacy endpoints: |
|---|---|
| | Fat thickness measurements using Ultrasound device |
| | 2. Fat thickness measurements using Caliper |
| | 3. Circumference measurements of the abdominal area using Measuring Tape |
| | 4. Investigator satisfaction using a pre-defined scale |
| | 5. Subject improvement and satisfaction using a pre-defined scale |
| | 6. Photography |
| Safety Endpoints | The number, severity and type of any adverse event recorded throughout the study and post treatment (immediate and delayed response) |
| Statistical | Descriptive statistics will be used to present changes in the assessments along the study |
| Methods | course. Circumference measurements and subject assessments' and satisfaction data will be |
| | analyzed using two-tailed Wilcoxon Signed Rank test and/or paired t-test (alpha=0.05) to |
| | analyze the data difference from baseline and longitudinal change. |

#### INTRODUCTION AND RATIONALE

# **Background**

Adipose tissue is a loose type of connective tissue specialized to store lipids. The majority of lipids stored in adipose cells are triglycerides formed from imported free fatty acids and glycerol. It is not uniformly distributed in the body. The major adipose depot is subcutaneous (about 80% of all body fat).<sup>1</sup> In men it normally represents 15-20% of body weight and in women, 20-25% of body weight. A certain amount of body fat is necessary for normal female reproduction and health. Subcutaneous adipose tissue helps to shape, cushion and insulate the body and provides padding to some organs.

Liposuction is a procedure that can help sculpt the body by removing unwanted fat from specific areas.<sup>2,3,4</sup> The increasing popularity of this procedure is associated with the evolution of techniques and equipment for fat removal, body reshaping and cellulite treatments. Besides the traditional suction-assisted lipoplasty, other options include ultrasound-assisted and external ultrasound-assisted liposuction, power-assisted liposuction, laser lipolysis as well as low-level laser-assisted liposculpture.<sup>5</sup>



| Clinical Study to Evaluate the Safety and Efficacy of the SlimShape Device for Abdominal Fat |
|---|
| and Circumference Reduction |

| Protocol # | DHF22621 | Rev. Date | October 8, 2017 | Page <b>9</b> of <b>39</b> |
|---|---|---|---|---|

The efforts in the search for alternative non-invasive or minimally invasive techniques and new tools aim mainly at reducing downtime, and facilitating treatment for reduction of the localized fatty tissue areas.<sup>6</sup>

The SlimShape device is a non-invasive, body countering system based on radiofrequency (RF) and vacuum energies. The SlimShape provide a non-invasive approach to achieve a desired aesthetic effect (reduction in abdominal fat and circumference). The system is designed to enable an automatic, hands-free, full abdominal treatment that is based on a predefined user protocol. In addition, the system incorporates a skin-temperature control into the protocol, enabling accurate, stable and safer treatment.

## **Device Descriptions**

## Syneron SlimShape Device

The SlimShape system is comprised of two main parts:

- The SlimShape console which houses the system's computer, control panel, electronics, discomfort button, cooling system and other power and control devices which operate and control the system.
- The SlimShape Applicator Belt incorporates an array of vacuum cavities; each cavity
  includes a pair of RF electrodes and a suction pad. Each of the cavities moves
  independently of the others, applying software-controlled vacuum and RF pulses in turn.

#### Main Console

The SlimShape console (Figure 1) incorporates the major modules required to deliver RF energy and negative air pressure (vacuum) to the applicator belt assembly, such as:

- RF generator
- Vacuum pump
- Computer
- 15" LCD control panel with touch-screen technology



Clinical Study to Evaluate the Safety and Efficacy of the SlimShape Device for Abdominal Fat and Circumference Reduction

 Protocol #
 DHF22621
 Rev. Date
 October 8, 2017
 



Figure 1: SlimShape System

#### The Applicator

The *SlimShape applicator Belt* (Figure 2) incorporates a linear array of vacuum cavities; each cavity includes a pair of RF electrodes and a suction pad. Each cavity has sufficient mechanical degrees of freedom with respect to the neighboring ones, so that when the applicator belt is attached to the patient it conforms to the body curvature. The SlimShape applicator is tightened to the skin, ensuring vacuum tightness by a strap and buckle mechanism. An array of vacuum, air and RF valves/switches will distribute the RF and vacuum energies sequentially between the cavities according to a software-controlled routine. Each cavity has temperature sensors that enable accurate control of the skin's temperature.



Figure 2: SlimShape Applicator



| Clinical Study to Evaluate the Safety and Efficacy of the SlimShape Device for Abdominal Fat |
|---|
| and Circumference Reduction |

| Protocol # | DHF22621 | Rev. Date | October 8, 2017 | Page <b>11</b> of <b>39</b> |
|---|---|---|---|---|
| Protocol # | DHF22621 | Rev. Date | October 8, 2017 | Page <b>11</b> of <b>39</b> |

A control button (Figure 3) is available to the patient in order to cease treatment if any discomfort is felt during the treatment. The discomfort button is designed to be held in the patient's hand during the entire treatment session. The patient should be instructed to press the button at any time he/she feels discomfort related to the treatment; this action stops the pulsing of vacuum and RF energy. The operator may then adjust the parameters or end the treatment session.



Figure 3: Discomfort Button

SlimShape is an upgraded version of the VelaShape device that is intended for abdominal fat reduction. The VelaShape device is cleared by the Food and Drug Administration (FDA). The upgraded version, the SlimShape device, is investigational and not yet FDA cleared.

#### STUDY DESIGN OVERVIEW

This study is a prospective, baseline controlled, multi-center, one arm clinical study showing the performance and safety of the SlimShape treatment for abdominal non-invasive fat and circumference reduction.

Up to 120 Healthy subjects in up to 10 investigational sites will be enrolled in this study. All subjects will undergo an assessment of their general health. During the treatment period, subject's fat thickness and circumference will be measured and up to three successive bi-weekly (two weeks interval) treatments will be performed.

The study subjects will undergo treatments with SlimShape device utilizing the SlimShape Applicator Belt.

During the follow-up period visit will be conducted as follow: 4 weeks (4wk FU), 8 weeks (8wk FU) and 12 weeks (12wk FU) post last treatment. Subject's fat thickness will be measured using 2 different methods (Calibrated Caliper and Ultrasound Imaging (USI)) and fat reduction will be assessed at each post baseline visit. Circumference will be measured in 3 measurements heights and circumference reduction will be assessed at each post baseline visit. Additionally, investigator and subject questionnaires will be completed. Finally, photography will be performed under visible light conditions of the front, right, left and back view. Most of the assessments will occur at each of the visits to the clinic.



| Clinical Study to Evaluate the Safety and Efficacy of the SlimShape Device for Abdominal Fat |
|---|
| and Circumference Reduction |

| Protocol # DHF22621 Re | v. Date October 8, 2017 | Page <b>12</b> of <b>39</b> |
|---|---|---|
|---|---|---|

#### **SUTDY OBJECTIVE**

The objective of this trial is to evaluate the safety and efficacy of the SlimShape device utilizing the SlimShape Applicator Belt for abdominal non-invasive fat and circumference reduction

## **Primary Objective**

Statistically significant abdominal fat reduction as measured by Ultrasound Imaging device post SlimShape treatments at 12 weeks follow-up (12wk FU) versus baseline.

# **Primary Safety Objective**

Evaluate the safety of the treatment with the SlimShape device utilizing the SlimShape Applicator Belt during all study.

## **Secondary Objectives**

- 1. Statistically significant abdominal fat reduction post SlimShape treatments as measured by USI device at Pre Tx.3, 4 weeks, and 8 weeks follow-up (4wk FU and 8wk FU) versus baseline.
- 2. Statistically significant abdominal fat reduction post SlimShape treatments as measured by Calibrated Caliper device at Pre Tx.3, 4 weeks, and 8 weeks follow-up (4wk FU and 8wk FU) versus baseline.
- 3. Statistically significant abdominal circumference reduction post SlimShape treatment/s at Pre Tx.2, Pre Tx.3, 4 weeks, 8 weeks and 12 weeks follow-up (4wk FU, 8wk FU and 12wk FU) versus baseline.
- 4. Investigator satisfaction:
  - Satisfaction assessment will be performed by the study investigator using a pre-defined scale questionnaire. The investigator will answer this questionnaire at each follow-up visit (4wk FU, 8wk FU and 12wk FU).
- 5. Subject improvement and satisfaction:
  Improvement and satisfaction assessment will be performed independently by the subject using a pre-defined scale questionnaire. The subjects will answer this questionnaire at each follow-up visit (4wk FU, 8wk FU and 12wk FU).

#### **Primary and Secondary Efficacy Endpoint**

Primary and secondary objectives will be measured using the next efficacy endpoints:

1. Fat thickness measurements using Ultrasound device



**Confidential** 

- 2. Fat thickness measurements using Calibrated Caliper device
- 3. Circumference measurements of the abdominal area using Measuring Tape
- 4. Investigator satisfaction using a pre-defined scale
- 5. Subject improvement and satisfaction using a pre-defined scale
- 6. Photography

## **Primary Safety Endpoint**

The number, severity and type of any adverse event recorded throughout the study and post treatment (discomfort (pain), immediate and delayed response).

- 1. Occurrence of expected post treatment immediate response including erythema and edema and during all study period based on predefined scale (Table 4).
- 2. Number, severity and type of any adverse event recorded throughout the course of the study.

#### STUDY POPULATION

## **Number of Subjects**

This study will be comprised of up to 120 subjects in up to ten (10) investigational sites. Subjects who meet all the inclusion and none of the exclusion criteria will be enroll.

## **Subject Withdrawal and Replacement**

Subjects enrolled in the study can discontinue their participation at any time for any reason without prejudice or reduction in the quality of their medical care. The investigators or sponsor can terminate a subject's participation in this study to protect the subject's health or if the subject fails to follow directions resulting in noncompliance to study procedures. Subjects who withdraw or are terminated from the study may be replaced to ensure at least 120 subjects have completed the study. Subjects who fail to complete the treatment will be replaced and will not be evaluable.

### **Inclusion Criteria**

A subject is eligible to participate in the study if he/she meets all the following inclusion criteria:

- 1. Signed informed consent to participate in the study.
- 2. Female and male subjects,  $\geq$  18 and  $\leq$  60 years of age at the time of enrolment
- 3. Fitzpatrick Skin Type I to VI
- 4. BMI interval:  $18.5 \le BMI \le 30$  (normal to overweight, but not obese).
- 5. If female, not pregnant, lactating and must be either post-menopausal, surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to

Clinical Study to Evaluate the Safety and Efficacy of the SlimShape Device for Abdominal Fat and Circumference Reduction

| Protocol # | DHF22621 | Rev. Date | October 8, 2017 | Page <b>14</b> of <b>39</b> |
|---|---|---|---|---|
|---|---|---|---|---|

- enrollment (i.e., oral contraceptives, contraceptive implant, barrier methods with spermicide or abstinence).
- 6. In addition, negative urine pregnancy test as tested before each treatment and at the last visit for women with childbearing potential (e.g. not menopause).
- 7. General good health confirmed by medical history and skin examination of the treated area.
- 8. Willing to follow the treatment and follow-up schedule and post-treatment care instructions.
- 9. Willing to refrain from a change in diet/ exercise/medication regimen for the entire course of the study.
- 10. Willing to have photographs and images taken of the treated areas to be used deidentified in evaluations, publications and presentations.

## **Exclusion Criteria**

A subject is not eligible for participation in this study if he/she meets any of the following exclusion criteria:

- 1. History of hypertension, ischemic heart disease, valvular heart disease, congestive heart failure, pacemaker/defibrillator, abdominal aortic aneurism
- 2. Current hyperlipidemia, diabetes mellitus, hepatitis, liver disease, HIV positive status, blood coagulopathy or excessive bleeding, autoimmune or connective tissue disease
- 3. Having or undergoing any form of treatment for active cancer, or having a history of skin cancer or any other cancer in the areas to be treated, including presence of malignant or pre-malignant pigmented lesions
- 4. Having any active electrical implant anywhere in the body, such as a pacemaker or an internal defibrillator
- 5. Having a permanent implant in the treated area, such as metal plates or an injected chemical substance such as silicone
- 6. Having undergone any other surgery in the treated areas within 12 months of treatment or during the study, including liposuction
- 7. Previous body contouring procedures in the treatment area within 12 months
- 8. History of skin disease in the treatment area, known tendency to form keloids or poor wound healing
- 9. History of epidermal or dermal disorders (particularly if involving collagen or microvascularity)
- 10. Suffering from significant skin conditions in the treated areas or inflammatory skin conditions, including, but not limited to, open lacerations or abrasions and active cold



Clinical Study to Evaluate the Safety and Efficacy of the SlimShape Device for Abdominal Fat and Circumference Reduction

| Protocol # DHF22621 Rev. Date October 8, 2017 | f <b>39</b> |
|---|---|
|---|---|

sores or herpes sores prior to treatment (duration of resolution as per the Investigator's discretion) or during the treatment course

- 11. Allergy to any component of the lotion (VelaSpray Ease) used in this study
- 12. Skin lesions in the treatment area other than simple nevi on physical examination (e.g., atypical nevus, tattoo, abrasions) including depressed scars in the treatment area
- 13. Very poor skin quality (i.e., severe laxity)
- 14. Abdominal wall diastasis or hernia on physical examination
- 15. Abnormal kidney, liver or coagulation functions, abnormal lipid profile or blood count within the last 3 months
- 16. Obesity (BMI > 30)
- 17. Childbirth within the last 12 months or breastfeeding women. Any acute or chronic condition which, in the opinion of the investigator, could interfere with the conduct of the study
- 18. Unstable weight within the last 6 months (i.e., ± 3% weight change in the prior six months)
- 19. Inability to comply with circumference measurement procedure (e.g., inability to hold breath for the required duration).
- 20. Participation in another clinical study involving same anatomical areas within the last 6 months (or 30 days in case different anatomical areas were treated in previous trial/s).
- 21. As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study.

#### **STUDY PROCEDURES**

## **Enrollment and Screening**

During the first visit, the research staff will screen the subject for eligibility to participate. The inclusion/exclusion criteria will be reviewed, the subject's medical history, an examination of the subject's skin in the treatment areas will be conducted.

The subject will review the informed consent form and the study will be explained to the subject including all risks, potential benefits, procedures, visit requirements, and other alternative treatment options. If the subject qualifies and wishes to participate they will complete the ICF with a signature and date. The original will be retained with subject's records and a copy will be provided to the subject.

The following measurements will be performed and recorded at the specified times throughout the study.

| SYNERON CANDELA | Clinical Study to Evaluate the Safety and Efficacy of the SlimShape Device for Abdominal Fat and Circumference Reduction | | | | |
|---|---|---|---|---|---|
| Syneron Medical Ltd.<br>Confidential | Protocol # | DHF22621 | Rev. Date | October 8, 2017 | Page <b>16</b> of <b>39</b> |

Table 2 – Clinical Evaluation Measurements and Tools

| Measurement | When to conduct | Method |
|---|---|---|
| Height | Baseline | Scale |
| Weight | Prior to all treatments (Tx.1, Tx.2 & | Scale |
| ВМІ | Tx.3), and at all follow-ups visits (4wk<br>FU, 8wk FU & 12wk FU) | Calculation |
| Fat thickness | Baseline, Prior to Tx.3, and at all | |
| UltraSound | follow-ups visits (4wk FU, 8wk FU & | Ultrasound device |
| measurements | 12wk FU) | |
| Fat thickness Caliper | | Calibrated Caliper |
| measurements | Prior to all treatments (Tx.1, Tx.2 & | cumprated camper |
| Circumference | Tx.3), and at all follow-ups visits (4wk | Standardized circumference measuring tape |
| measurements | FU, 8wk FU & 12wk FU). | |
| Photographs | | Standardized digital photographs |
| Urine pregnancy test | Prior to all treatments (Tx.1, Tx.2 & Tx.3), and at the last follow-up visit (12wk FU) | Urine pregnancy test |
| Immediate response assessment | Immediately after each treatment (Tx.1, Tx.2 & Tx.3) | Post Treatment Side Effect Severity Scale (Table 4) |
| Investigator satisfaction | At all follow-up visits (4wk FU, 8wk FU | Satisfaction Questionnaire (Table 6) |
| Subject satisfaction | and 12wk FU) | Satisfaction Questionnaire (Table 6) |
| Subject improvement assessment | | Improvement Questionnaire (Table 5) |
| Safety | During treatment and throughout study. | Examination of skin in the treated area, interview subjects, Adverse Events form, Occurrence and Severity Ratings, as well as relation to treatment, action taken and outcome |



Figure 4: Study Flow-Chart (Visits at the Clinic)



Clinical Study to Evaluate the Safety and Efficacy of the SlimShape Device for Abdominal Fat and Circumference Reduction

## **Pre-Treatment Procedures**

It is expected that the screening and baseline procedures will be conducted during the same visit as the treatment (prior to the treatment). The treatment visit procedures will take up to 1.5 hours.

## Screening

- ICF Prior to any study procedures, informed consent will be obtained. When the subject fully understands the possible benefits and risks of the study, the subject will be asked to sign and date the informed consent form (ICF). The subject will be given a copy of the signed ICF.
- 2. Subject ID subjects will be assigned a study subject ID number.
- 3. Medical History A medical history will be obtained to determine if the subject meets the study criteria, including a list of all prescribed and over the counter medications taken within the previous 6 months will be recorded.
- 4. Skin Exam The subject will undergo a routine skin exam to determine if they meet the study criteria including the presence of fatty tissue deposits in the treatment area.
- 5. BMI the volunteers' height and weight will be taken for calculation of BMI.
- 6. Pregnancy Screen Subjects who are capable of becoming pregnant will undergo a urine pregnancy test. This will be repeated prior to all treatments, and at the end of the study (last FU visit/ 12wk FU). If the Screening and Treatment procedures are not conducted on the same day, the urine pregnancy test will be repeated on the first treatment day.
- 7. Scheduling: Subjects will be scheduled to return for the baseline and first treatments visit within 14 days following the screening visit. It is preferable the baseline procedures and Tx.1 will be conducted immediately after the Screening visit.

#### **Baseline**

- 1. Photography Baseline photographs will be obtained using a consistent camera and subject placement settings with a digital imaging system.
- 2. BMI the subject weight and height will be taken if baseline visit occurs on a different day than the screening visit.



| Clinical Study to Evaluate the Safety and Efficacy of the SlimShape Device for Abdominal Fat |
|---|
| and Circumference Reduction |

| Protocol # DHF22621 Rev. Date October 8, 2017 | Page <b>18</b> of <b>39</b> |
|-----------------------------------------------|-----------------------------|
|-----------------------------------------------|-----------------------------|

#### Measurements

## Measure the Fat Thickness at the Treated Area – Calibrated Caliper

Assess fat thickness at treatment area prior starting the treatment using calibrated caliper.

## Measure the Fat Thickness at the Treated Area – Ultrasound Imaging Device

Ultrasound Imaging (USI) provides a valid way for measuring fat thickness using known interfaces observed in any individual. USI is relies on the ability to recognize different sub-skin interfaces and correctly identifying them, such as the **dermis** and the **subcutaneous fat layer** interfaces.

- a) Treated area is defined below the sternum and above the iliac. Mark the rectangle of the treated area with white pencil.
- b) Measure 2-4 cm from each edge of the umbilicus (superiorly and inferiorly) and 1.5-3 cm medially and laterally from the ends of these points (as illustrated in Figure 5, white lines). Make sure that the measurement points selected are at least 1 cm from the edges of the treatment area (including the width of the USI transducer, see green arrows in Figure 5).



UR-Upper Right measurement point, UL-Upper Left measurement point, LR-Lower Right measurement point, LL-Lower Left measurement point

Figure 5: Ultrasound Measurements Points

c) Mark the treated area and the measurements points on the transparency, to ensure measurement of the same point in each subsequent visit.

| SYNERON CANDELA | Clinical Study to Evaluate the Safety and Efficacy of the SlimShape Device for Abdominal Fat and Circumference Reduction | | | | |
|---|---|---|---|---|---|
| Syneron Medical Ltd.<br>Confidential | Protocol # | DHF22621 | Rev. Date | October 8, 2017 | Page <b>19</b> of <b>39</b> |

- d) Ultrasound measurements should be obtained from the edges of the measurement points, laterally (see **Figure 5 above, yellow dashed lines**).
- e) Place the applicator on the skin surface at angle of 90° (located the applicator under the measurement point line for consistency).
- f) Measurement should include all the area between the dermis and end of the fat tissue fascia. At least 2 measurements should be done in each measurement point.

#### Marking height of circumference measurement

The abdominal circumference measurement will be marked at **1cm Above Iliac Height** (middle height of the treated area circumference). Patient should stand up straight when arms are placed at the rear of neck and head is positioned towards the horizon (Figure 7). Elbows will be positioned in front of the body (Figure 7).

The height for the circumference measurement will be marked at the anterior abdomen, at the back and at each lateral side of the body. Additional measurements will be taken at: **Waist Height** (upper height of the treated area circumference) and at **1.5inch** (**3.81cm**) **Below Navel Height** (lower height of the treated area circumference) See Figure 6 below.









Figure 7: Body poisoning during marking height for circumference measurement

The 1cm Above Iliac Height, Waist Height and 1.5inch (3.81cm) Below Navel Height will be measured using the height measuring device (supplied by Syneron Medical). The marking pencil will be placed horizontally at the stage of the measurement device during the marking procedure. (Figure 7)

Height of all measurements point will be recorded in the CRF (will used as reference for the next visits measurements). As well, the circumference results of each height will be recorded at each visit.

### <u>Measuring Circumference</u>

Abdominal circumference is measured to quantify the treatment effect. This procedure will be performed and recorded every visit at the clinic, immediately following the measurement of height marking.

In order to achieve reproducible measurement results, the following requirements should be fulfilled:

- 1. Patient should be wearing underwear and barefoot during circumference measurement.
- 2. Patient should stand up straight when arms are placed at the rear of neck and head is positioned towards the horizon. Elbows will be positioned in front of the body (see Figure 8A).
- 3. The measurement tape (supplied by Syneron Medical) should be in parallel to the floor during the measurement (see Figure 8B).
- 4. The circumference measurement tape should be placed <u>under</u> the marked reference points, in order to maintain repetitive height of the measurement.

| SYNERON © CANDELA | Clinical Study to Evaluate the Safety and Efficacy of the SlimShape Device for Abdominal Fat and Circumference Reduction | | | | |
|---|---|---|---|---|---|
| Syneron Medical Ltd.<br>Confidential | Protocol # | DHF22621 | Rev. Date | October 8, 2017 | Page <b>21</b> of <b>39</b> |

 Middle measurement should be taken at the level of the <u>1cm Above Iliac Height</u>. Additional two circumference measurements at <u>Waist Height</u> and <u>1.5inch (3.81cm)</u> <u>Below Navel Height</u> will be taken. This height levels should be recorded for follow up assessments.

6. Consecutive measurements should be performed at the same height recorded at baseline. In order to assure that the measuring tape is parallel to the floor, several reference points should be marked around the treatment area and the measuring tape should be placed such that it is aligned with them.



Figure 8: Patient positioning during circumference measurements (A) and measuring device position around the abdomen (B)

- 7. The measurement device should be activated at a constant tension to achieve an exact measure of the circumference (use measurement device supplied by Syneron only).
- 8. In order to minimize measurement inaccuracies originating from human error, it is recommended that, whenever possible, the same operator re-measures the patient at approximately at the same hour of day (± 3 hours).
- 9. Patients should be under fasting for at least 3 hours prior to circumference measurement.

#### **Treatment Procedure**

Subjects will receive treatments with SlimShape device utilizing the SlimShape Applicator Belt on the anterior abdomen.

Prior to each treatment measurements of weight, fat thickness (by Caliper & Ultrasound), and abdominal circumference will be done according to the references from the enrollment visit



Clinical Study to Evaluate the Safety and Efficacy of the SlimShape Device for Abdominal Fat and Circumference Reduction

 Protocol #
 DHF22621
 Rev. Date
 October 8, 2017
 

(Baseline/ prior to Tx.1). Only patients who are eligible for treatment will be allowed to undergo the SlimShape procedure.

Enrolled subjects will undergo up to 3 successive (according to investigator decision) bi-weekly (2 weeks interval) treatments (Tx.1, Tx.2 and Tx.3). Additional three (3) visits in the clinic will be occurred to follow-up the abdominal fat and circumference reduction at visits 4, 5 and 6 (4 weeks, 8 weeks and 12 weeks following last treatment).

### **SlimShape Treatment Procedure**

#### **General Treatment Instructions**

- 1. Place the patient so that he/she is lying on his/her back, with the legs extended. In this position, the abdomen is fully accessible and treatment can be easily performed.
- 2. Remove any jewelry in the area of the application site.
- 3. Ensure that the subject skin in the entire treatment is clean. The skin should be cleaned with water and soap and hairs that exist in the treatment areas will be shaved.
- 4. Ensure that the applicator belt is clean or wipe with 70% alcohol and allowed to dry.
- 5. The choice of treatment settings should take into consideration not only the severity of the treated condition (fat layer), but also the subject's skin type, tendency to bruise, the specific anatomical location (abdomen), and comfort.
- 6. Immediately prior the treatment, apply a generous amount of the commercial VelaEase treatment lotion, RF coupling lotion. You may need to re-apply the lotion if required.
- 7. Position the SlimShape Applicator Belt at the correct/ chosen treatment area (on the abdomen).
- 8. There should be a complete seal between the applicator and the skin during the treatment session. If you hear air being sucked into the chamber, this indicates that the contact between the skin and the belt chambers is not ideal for vacuum creation. This usually means that the applicator is not positioned properly at that moment, which tends to happen in curved or bony areas, so special attention is required when treating such areas. Changing the orientation of the applicator slightly may solve this problem.
- 9. The applicator belt chambers should have equal compression/contact with the skin to ensure safe and effective RF delivery.
- 10. Secure the magnetic pads on the sides of both belts, on both sides of the patient and tight the SlimShape belt.
- 11. Select the desired treatment protocol.

| SYNERON CANDELA | Clinical Study t | Clinical Study to Evaluate the Safety and Efficacy of the SlimShape Device for Abdominal Fat and Circumference Reduction | | | |
|---|---|---|---|---|---|
| Syneron Medical Ltd.<br>Confidential | Protocol # | DHF22621 | Rev. Date | October 8, 2017 | Page <b>23</b> of <b>39</b> |

- 12. Full operating procedure, software screens and parameters are described in the device user manuals and instruction will be provided prior to the start of the study.
- 13. Expected post treatment side effects are limited to Erythema (blanchable/non-blanchable), Edema, Heat sensation, Hematoma and Pain sensation.

| SYNERON © CANDELA | Clinical Study to Evaluate the Safety and Efficacy of the SlimShape Device for Abdominal Fat and Circumference Reduction | | | | |
|---|---|---|---|---|---|
| Syneron Medical Ltd.<br>Confidential | Protocol # | DHF22621 | Rev. Date | October 8, 2017 | Page <b>24</b> of <b>39</b> |

# **Post Treatment Procedures**

- 1. Safety aspect will be assessed before and after each treatment:
  - a. Clinical effects All visible and palpable immediate response will be recorded for the entire treatment area using a 4-point severity scale (Table 4)
  - b. Adverse Events Record the number, severity and type of any adverse event occurred before, through and after treatments.

## **Return Visits**

All subjects will be requested to return to the clinic at the following time-points during the study in order to assess the clinical performance of the device:

- Visit 4: FU1 4 weeks (±7 days) post last treatment.
- Visit 5: FU2 8 weeks (±7 days) post last treatment.
- Visit 6: FU3 12 weeks (±7 days) post last treatment.

At each return visit the following procedures will be conducted and data recorded:

- Weight.
- Ultrasound fat-thickness measurements.
- Caliper fat-thickness measurements.
- Circumference measurements.
- Skin assessment for clinical effects due the procedures:
  - Post treatment response and adverse events.
- Photographs as conducted at baseline.
- Satisfaction questionnaire performed by the investigator using the Global Aesthetic Improvement (GAI).
- Completion of the Subject Follow Up questionnaire:
  - Subjective Improvement and satisfaction performed by the subject using the Global Aesthetic Improvement (GAI).
- At the final visit a urine pregnancy test will be performed for women with childbearing potential.



| Clinical Study to Evaluate the Safety and Efficacy of the SlimShape Device for Abdominal Fat |
|---|
| and Circumference Reduction |

#### **DATA ANALYSIS**

## Recording

All data will be recorded on site source documents and transcribed onto Case Report Forms (CRFs). The site will be monitored by Syneron staff or designees to assure adherence to the clinical trial requirements, subject safety, protocol procedures, and for data accuracy. The Case Report Forms and images will be reviewed and retrieved during the monitoring visit. All source documentation will remain in the subject's files at the site.

Review and Analysis of all data collected will be conducted by the Sponsor or designee as described for this protocol with the following data:

### **Demography and Baseline Measurements**

Demographic and baseline/screening measurements (e.g., weight, height and digital images) will be collected and descriptively presented.

#### **Treatment Visit**

Skin assessment by the PI, photographs of the treated region, and pain scores will be collected used to document any adverse events to assess the device performance.

#### **Follow-up Visit Measurements**

Follow-up measurements for weight, circumference and digital images will be used for comparative measurements with their respective measurement at baseline. Primary endpoints will be evaluated 12 weeks post last treatment. Secondary endpoints may be evaluated at all visits.

#### Safety

Safety of device procedure will be evaluated through skin assessments by the PI and research staff. The occurrence and severity of all complications from the start of the study will be recoded.

## **Protocol Revisions and/or Deviations**

With the exception of emergency situations, no changes or deviations in the conduct of this protocol will be permitted without the prior approval of the sponsor.

The IRB/IEC that granted original approval for the study must be notified of all changes in the protocol, and will approve any change or deviation that may increase risk to the subject, and/or that may adversely affect the rights of the subject or validity of the investigation.



| Clinical Study to Evaluate the Safety and Efficacy of the SlimShape Device for Abdominal Fat |
|---|
| and Circumference Reduction |

| Protocol # DHF22621 Rev. Date October 8, 2017 Page 26 of 3 |
|------------------------------------------------------------|
|------------------------------------------------------------|

In the event of an emergency, the Investigator will institute any medical procedures deemed appropriate. However, all such procedures must be promptly reported to the sponsor and the IRB/IEC.

## **ADVERSE EVENTS (AE)**

An adverse event (AE) is any adverse change in health or side effect that occurs in a study participant during their participation in the study.

## **Anticipated Adverse Effects**

Following treatment with the <u>SlimShape</u> the following local adverse effects could occur (anticipated):

Purpura
Erosion

Blister
Pain/soreness

➤ Bruising ➤ First degree burn

BullaeSecond degree burn

An adverse event (AE) is any undesired clinical occurrence in a study subject as indicated by signs, symptoms, illnesses, events that develop or worsen in severity in association with the study when deemed by the Investigator to be related to use of the device or study procedures. The Investigator will document all adverse signs and symptoms regardless of severity or frequency that are either volunteered by subjects or observed during the course of the study that are related to the device. The Investigator will also record adverse experiences of subjects resulting from concurrent illnesses, reactions to concurrent medications, or progression of disease states that the Investigator deems related to the device. Included in the description will be the nature of the sign or symptom, the date of onset, whether the event was serious, the severity, the relationship to study procedures or investigational device, the action taken, the date of resolution, and the outcome. The Principal Investigator will determine the relationship of the adverse device effect to the investigational device.

## **Unanticipated Adverse Device Effects**

For device studies, part 21 CRF 812.3(s) uses the term unanticipated adverse device effect which is defined as any serious adverse effect on health or safety or any life-threatening problem or death caused by, or associated with the device, if that effect, problem, or death was not previously identified in nature, severity, or degree of incidence in the investigational plan or application (including a supplementary plan or application), or any other unanticipated serious problem associated with a device that relates to the rights, safety, or welfare of subjects.



# Clinical Study to Evaluate the Safety and Efficacy of the SlimShape Device for Abdominal Fat and Circumference Reduction

 Protocol #
 DHF22621
 Rev. Date
 October 8, 2017
 

Significant device failure may constitute an adverse event if an undesirable experience occurs. This definition includes any event resulting from insufficiencies or inadequacies in the instructions for use or the deployment of the device, or any event that is a result of a user error.

## All unanticipated adverse effects will be graded as follows:

Mild: Sign or symptom, usually transient, non-life-threatening requiring no special

treatment and generally not interfering with usual activities.

Moderate: Sign or symptom, non-life-threatening which may be ameliorated by simple

therapeutic measures, and may interfere with usual activity.

Major: Sign or symptom that is intense or debilitating but non-life-threatening and

that interferes with usual activities. Recovery is usually aided by therapeutic measures and the discontinuation of the study device may be required.

Severe: Any untoward medical occurrence that at any time results in death or life-

threatening illness, resulting in persistent or significant disability/incapacity.

The relationship of the adverse effect to the study is defined as follows:

**Probable:** An adverse event has a strong temporal relationship to study device, and

another etiology is unlikely or significantly less likely.

**Possible:** An adverse event has a strong temporal relationship to the study device, and

an alternative etiology is equally or less likely compared to the potential

relationship to study device.

**Probably not:** An adverse event has little or no temporal relationship to the study device

and/or a more likely alternative etiology exists.

**Not related:** An adverse event has no temporal relationship to study device or has a much

more likely alternative etiology.

## Reporting Adverse Events (AE) and Serious Adverse Events (SAE)

**Anticipated Adverse Events:** Anticipated adverse events in this study include Purpura, blistering, bruising, bullae, erosion, soreness and burn. If an unanticipated adverse event occurs at any time during or after the use of the SlimShape device, the Investigator must report it to Syneron.

The Investigator must report all unanticipated adverse device effects that are serious in nature to the clinical study monitor immediately or within twenty-four hours by telephone (see below). If such an unanticipated adverse device effect is reported after normal working hours, the Investigator will leave a voice message at the monitor's telephone number with accompanying report of the unanticipated adverse device effect faxed or sent to the fax number/e-mail address below:



# Clinical Study to Evaluate the Safety and Efficacy of the SlimShape Device for Abdominal Fat and Circumference Reduction

Protocol # DHF22621 Rev. Date October 8, 2017 

Ruthie Amir, MD, Global VP of Clinical Affairs

Telephone/Fax No.: From the U.S. 011 (972) 73-244-2349

011 (972) 54-300-3164 (cell)

E-mail: ruthiea@syneron.com

A written report prepared by the Principal Investigator must follow within five working days to both the IRB and to Syneron and should include a full description of the event and sequence.

## Measures taken to protect the rights and welfare of subject

Research records will be available to study personnel, the sponsor, Ethics Review Committee and regulatory agencies as required. Research records may be used for purposes of medical education, after removal of subject names or other identifying information. In the ICF the subjects will be informed that the photographs and video taken of them during the study may be made available to the sponsor for marketing and instructional purposes, after removal of identifying information. All images collected will be stored without personal subject identifiers at the site and at Syneron.

# **RISK/BENEFIT ANALYSIS**

#### Risks

Syneron has determined that the *SlimShape* system is non-significant risk device. As indicated in the AE section, the anticipated risks associated with the use of both of the systems are:

Purpura
Erosion

Blister
 Bruising
 Bullae
 Pain/ soreness
 First degree burn
 Second degree burn

Over 2500 subjects worldwide participated in clinical research and underwent treatment with the different *VelaShape family* devices. The *SlimShape* device will be used in this study was previously used in studies and emitted the same acoustic energy. To date, no serious adverse events or unanticipated AEs have been reported. The reported AEs relate to skin and subcutaneous tissue, confined to the treatment area and were all mild in nature and resolved within the study period.

# Potential benefits to participating individuals and to society

Subjects may or may not benefit from reduction of subcutaneous fatty tissue on the treated area via a non-invasive technique resulting in body contouring improvement. All subjects in the treatment groups are expected to have some benefit from the treatment procedures as would



| Clinical Study to Evaluate the Safety and Efficacy of the SlimShape Device for Abdominal Fat |
|---|
| and Circumference Reduction |

| Protocol # | DHF22621 | Rev. Date | October 8, 2017 | Page <b>29</b> of <b>39</b> |
|---|---|---|---|---|
|---|---|---|---|---|

be expected for the commercial devices (*SlimShape*). Subject will receive all treatment procedures at no cost. This study will benefit the advancement of medicine by generating data on safety and efficacy that will aid in the development of an alternative treatment options to procedures with higher potential risks subjects, such as liposuction. The results of this study will help to determine whether this device is safe and effective for improvement of localized subcutaneous fat.

### **Conclusion:**

In light of the potential benefits of non-invasive body contouring relative to its risks, the potential benefits associated with the use of the SlimShape System outweigh its risks, supporting study initiation.

#### ETHICS AND GOOD CLINICAL PRACTICE

This study will be carried out in compliance with the following:

- Syneron Standard Operating Procedures.
- Declaration of Helsinki, concerning medical research in humans (Recommendations Guiding Physicians in Biomedical Research Involving Human Subjects, Helsinki 1964, amended Tokyo, 1975, Venice 1983, and Hong Kong 1989).
- US Code of Federal Regulations (Title 21CFR including parts 50, 56 and 812 governing informed consent and IRB regulations).
- International Conference on Harmonization (ICH) Harmonized Tripartite Guideline for Good Clinical Practice (GCP), 1996.

#### **QUALITY ASSURANCE AND STUDY MONITORING**

## Study Monitoring/Auditing/Inspection

The Study Monitor will be responsible for monitoring the study sites to review the data being collected. The sponsor shall implement and maintain quality control and quality assurance procedures with written standard operating procedures (SOPs) to ensure that the trial is being conducted and data are generated, documented and reported in compliance with the protocol, Good Clinical Practice (GCP) and applicable regulatory requirements. Visits will be made prior to the initiation of the study, at scheduled intervals throughout the study, and at termination of the study.

Once enrollment and treatments have begun, monitoring visits will take place more frequently pending enrollment and study activities.



| Clinical Study to Evaluate the Safety and Efficacy of the SlimShape Device for Abdominal Fat |
|---|
| and Circumference Reduction |

| Protocol # | DHF22621 | Rev. Date | October 8, 2017 | Page <b>30</b> of <b>39</b> |
|---|---|---|---|---|
|---|---|---|---|---|

The sponsor and site will maintain regular phone and e-mail correspondence throughout the study to confirm compliance of study procedures.

The investigator/institution agrees to allow the monitor and other authorized personnel direct access to source data/ documents for trial related monitoring, the clinical supplies storage/dispensing area and to provide all documents in the Investigator Regulatory Binder for review, and to assist site auditors in their activities if requested. Requests by the Health Canada or regulatory agencies of other countries to inspect the study site may be made after adequate notification. The investigator may be required to assist the regulatory inspectors in their duties, if requested.

#### ADMINISTRATIVE PROCEDURES

## **Supply and Disposition of Study Device**

The *SlimShape* device and VelaEase (coupler agents) will be supplied to the participating clinic. The device will be maintained by the Sponsor, as needed. Unused equipment or coupler agents will be returned to the sponsor at the end of the study. At the end of all planned treatment sessions the devices will be returned to Syneron.

## **Control & Disposition of the Investigational Device**

The *SlimShape* device will be used according to the instructions of the Sponsor and manufacturer, Syneron Medical. At the end of this study, any materials provided specifically for use in this study may be returned to the Sponsor, as described in the Clinical Trial Agreement and study budget.

## <u>Informed Consent</u>

The Study Personnel will obtain written Informed Consent prior to the subject's participation in any study procedures. The Study Personnel will inform the subjects of the experimental procedure to be utilized and assure the subjects that their decision regarding participation in the study will have no bearing on the quality of medical care received and that their decision whether to participate in the study is strictly voluntary.

During the initial interview, the subject will be assured that they are free to change their mind and will be allowed to participate in the study or withdraw from the study with no adverse effect on their standard medical care.



| Clinical Study to Evaluate the Safety and Efficacy of the SlimShape Device for Abdominal Fat |
|---|
| and Circumference Reduction |

| Protocol # DHF22621 Rev. Date October 8, 2017 | Protocol # |
|---|---|
|---|---|

### **Monitoring Plan**

At least 3 monitoring visits are projected during the whole study. The frequency of which will be based on enrolment, study activities and the study visit scheduled. The first visit is scheduled at the initiation of the study prior to the first subject treatment in the study. The second visit is scheduled after enrolment and treatment has been initiated and a third visit will be for a close-out visit for the study. Interim visits may be conducted as needed to assure compliance to the study protocol and regulatory requirements. The number and frequency of monitoring visits may also be increased per the sponsor decision to collect data and images post treatment.

## **Case Report Forms**

Paper case report forms will be used in this trial. All protocol-required information collected during the study must be entered in the appropriate field of the case report form (CRF). The investigator, or designated representative, should complete the appropriate CRF fields as soon as possible after information is collected. The information must match the information that exists as source documents in the clinic chart, hospital chart, and/or investigator's files. An explanation should be given for all missing data.

It is the investigator's responsibility to assure the accurate completion, review, and approval of all CRFs and the timely completion and submission of all adverse event forms.

### **Record Maintenance**

The investigator shall retain a copy of all study documents in accordance with the FDA regulations which specify that records should be kept for a period of two years: 1) following the date a marketing application either is approved or disapproved for the use, or 2) following notification to FDA that no application is being filed and/or that the study has been discontinued.

If an investigator leaves the study site before record retention obligations have expired, the sponsor should be notified in writing of the person designated to retain the study documents during and after the study.

Handling of clinical data. The data are entered into a secure database that only the sponsor has access to. Admission to the database requires access to a password-protected network secured by the Sponsor. This database is maintained by Syneron that performs backups, data verification, and application upgrades. All equipment housing the clinical data is located in locked rooms or a secure computer network. The only individuals, who view, extract and analyze data for protocol reports and publications are physicians and nurses who are members of the study team or Sponsors. Only authorized personnel of the Sponsors have access to databases.

Any paper copies of subject medical records or research records are stored in secure cabinets at the study site.



| Clinical Study to Evaluate the Safety and Efficacy of the SlimShape Device for Abdominal Fat |
|---|
| and Circumference Reduction |

| Protocol # | DHF22621 | Rev. Date | October 8, 2017 | Page <b>32</b> of <b>39</b> |
|---|---|---|---|---|

### **PUBLICATION POLICY**

The investigator will not publish the study results and will not disclose confidential information received from Syneron without prior written agreement from Syneron. Such confidential information shall include any and all information relating to this study as described in the Clinical Trial Agreement. In the event that Syneron consents to the publication of data from this study, the investigator will provide Syneron manuscripts for review thirty days before submission for publication. Syneron will have no editorial rights over manuscripts. The investigator will also provide Syneron with advance notice of at least (30) days, of any presentation, lecture, abstract session, etc., in which any results from the study will be disclosed.



| Clinical Study to Evaluate the Safety and Efficacy of the SlimShape Device for Abdominal Fat |
|---|
| and Circumference Reduction |

| Protocol # DHF22621 Rev. Date October 8, 2017 Page 33 of 3 |
|------------------------------------------------------------|
|------------------------------------------------------------|

#### **BIBLIOGRAPHY**

- 1. Arner P. *OBESITY AND THE ADIPOCYTE, Regional adipocity in man*. Journal of Endocrinology (1997) 155, 191–192
- 2. Illouz YG, de Villiers YT. *Body Sculpturing by Lipoplasty*. Edinburgh: Churchill Livingstone, 1989.
- 3. Gasparotti M. Superficial liposuction: a new application of the technique for aged and flaccid skin. Aesthet Plast Surg (1992) 16, 141–53
- 4. Adamo C, Mazzocchi M, Rossi A and Scuderi N. *Ultrasonic liposculpturing. extrapolations* from the analysis of in vivo sonicated adipose tissue. Plast Reconstr Surg (1997) 100, 220–6
- 5. Goldman A. *Submental Nd:YAG Laser-Assisted Liposuction*. Lasers in Surgery and Medicine 38:181–184 (2006).
- 6. Hexsel D, Serra M, Mazzuco R, Dal'Forno T, Zechmeister D. *Phosphatidylcholine in the treatment of localized fat.* J. Drugs Dermatol. 2003 Oct;2(5):511-8.

| SYNERON © CANDELA' | Clinical Study to Evaluate the Safety and Efficacy of the SlimShape Device for Abdominand Circumference Reduction | | |
|---|---|---|---|
| Syneron Medical Ltd. Confidential Protocol # DHF22621 Rev. Date October 8, 2017 | | October 8, 2017 | Page <b>34</b> of <b>39</b> |

# **APPENDIX I – STUDY SUMMERY**

| | Screen /<br>Baseline*<br>Tx.1 | Tx.2<br>2 weeks ± 5<br>days | Tx.3<br>2 weeks ±<br>5 days | 4 weeks<br>Follow-Up<br>(4wk FU)<br>±7 days | 8 weeks<br>Follow-Up<br>(8wk FU)<br>±7 days | 12 weeks<br>Follow-Up<br>(12wk FU)<br>±7 days |
|---|---|---|---|---|---|---|
| Informed Consent<br>Process | X | | | | | |



Clinical Study to Evaluate the Safety and Efficacy of the SlimShape Device for Abdominal Fat and Circumference Reduction

Syneron Medical Ltd. Confidential

Protocol # DHF22621 Rev. Date October 8, 2017 

| Eligik | oility Screening & | | | | | | |
|--------------------------|--------------------|---|---|---|---|---|---|
| | cal History | Х | | | | | |
| | Photography | X | X | Χ | X | Χ | Χ |
| | Height | X | | | | | |
| N | Weight (BMI | Х | Х | Х | Х | Х | Х |
| ME | calculation) | ^ | ^ | ^ | ^ | | |
| ATI | Transplant | x | | | | | |
| 'RE | Preparation | | | | | | |
| PERFORM BEFORE TREATMENT | Fat Thickness | | | | | | |
| <u> </u> | Ultrasound | х | | X | X | X | x |
| BEI | Measurement | | | | | | , |
| Σ | (Prior Strapping) | | | | | | |
| OR | Fat Thickness | | | | | | |
| RF | Caliper | X | X | Х | X | X | X |
| PE | Measurement | | | | | | |
| | Circumference | X | Х | X | X | Х | х |
| | Measurements | Λ | Λ | ^ | A | Α | Λ |
| Treat | ment | X | X | X | | | |
| Safet | y Monitoring | X | X | Χ | X | X | X |
| Subje | ect Questionnaire | | | | X | Χ | X |
| Investigator | | | | | х | Х | Х |
| Questionnaire | | | | | ^ | ^ | ^ |
| Urine Pregnancy Test | | Х | Х | Х | | | Х |
| End of Participation | | | | | | | Х |
| (Termination) | | | | | | | ^ |

Clinical Study to Evaluate the Safety and Efficacy of the SlimShape Device for Abdominal Fat and Circumference Reduction

Protocol # DHF22621 Rev. Date October 8, 2017 

## **APPENDIX II - SCALES**

## <u>Table 4 - Post Treatment Side Effect Severity Scale</u>

| (0) Absent / None |
|-------------------|
| (1) Mild |
| (2) Moderate |
| (3) Severe |

# <u>Table 5 – Global Aesthetic Improvement (GAI) Scale</u>

| (3) Significant improvement |
|-----------------------------|
| (2) Moderate improvement |
| (1) Slight improvement |
| (0) No change |
| (-1) Slightly worse |
| (-2) Moderately worse |
| (-3) Significantly worse |

## <u>Table 6 – Satisfaction Scale</u>

| (2) Very satisfied |
|------------------------|
| (1) Satisfied |
| (0) No opinion |
| (-1) Dissatisfied |
| (-2) Very dissatisfied |



| Clinical Study to Evaluate the Safety and Efficacy of the SlimShape Device for Abdominal Fat |
|---|
| and Circumference Reduction |

#### **APPENDIX III - PHOTOGRAPHY**

At each of the specified time points; photographs of the treated areas should be taken by investigator or their designee.

- Photographs should be taken in a private room or area of the clinic under controlled conditions, including the distance from the camera to the subject, height of the camera, background, camera positioning, subject's positioning and lighting in order to achieve high-quality before & after sets.
- Consistent lighting- Lighting should be projected from about 45° angle in order to emphasize the body appearance.
- It is important to keep a constant distance between the subject's feet (use "sticky feet" or another way of marking) in order to properly present the effect of the treatment. The recommended distance between the feet is ~20 cm, but the main point is not to make this distance too small, so the thighs touch each other, or too large.
- The disposable underwear should be used for all photographs of all of the anatomical areas at all time points.
- For consistency purposes, the same person should ideally take all study photographs, especially per area and subject.
- The digital files should follow a consistent standard naming scheme containing subject initials and study ID #, visit or visit date.

## **Specific photography details:**

#### Abdomen:

Three photographs should be taken at each specified time point

- Front
- 45º from the right side
- 90º from the right side
- 45º from the left side
- 90º from the left side

The subject's arms should remain out of the way; it is best to either cross them over each other in front of the chest or hold them up at a 90° angle to the body, ensuring that they do not rest on the chest or touch the body and that they do not cast a shadow in the photograph.



Clinical Study to Evaluate the Safety and Efficacy of the SlimShape Device for Abdominal Fat and Circumference Reduction

| Protocol # | DHF22621 | Rev. Date | October 8, 2017 | Page <b>38</b> of <b>39</b> |
|---|---|---|---|---|
|---|---|---|---|---|

## **APPENDIX IV - CLINICAL TRIAL ACKNOWLEDGEMENT**

| outlined herein and in accordance wi<br>universal regulations pertaining to clinic | | cices, as well as with local and |
|---|---|---|
| Investigator's Signature | - | Date |
| Name | _ | |
| Clinic | _ | Street Address |
| City, State & Zip Code | _ | Country |
| Phone # | - | |
| Fax # | - | |
| E-mail Address | _ | |

I have read and understood the foregoing protocol, and agree to conduct this clinical study as

Clinical Study to Evaluate the Safety and Efficacy of the SlimShape Device for Abdominal Fat and Circumference Reduction

| Protocol # | DHF22621 | Rev. Date | October 8, 2017 | Page <b>39</b> of <b>39</b> |
|---|---|---|---|---|
| | | | , | J |